CLINICAL TRIAL: NCT00766701
Title: Pivotal Study for Assessment of Cervical Neoplasia Using Fluorescence and Reflectance Spectroscopy
Brief Title: Spectroscopic Evaluation of Cervical Neoplasia
Status: Completed | Type: Observational
Sponsor: Guided Therapeutics (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Dr. Lisa Flowers M.D., Emory University
Other Study IDs: GT1
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Last update posted 2008-10-06 (Estimated); Status verified 2008-10

CONDITIONS: Cervical Neoplasia
MeSH Terms: interventions — Spectrum Analysis; Quantitative Phase Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — histology slides
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Procedure: Spectroscopy and Digital Imaging — Procedure: Spectroscopy and Digital Imaging
  Other Names: Spectroscopy; Digital Imaging

SUMMARY:
The overall objective of this study is to evaluate whether fluorescence and reflectance spectroscopy can improve the ability to detect the presence of premalignant lesions on the cervix.

The specific aims of the study are:

* To compare information obtained from fluorescence and reflectance spectroscopic measurements of the cervix with standard methods for detecting cervical pre-cancers.
* To validate previously developed algorithms for discriminating between normal and pre-cancerous tissue based on spectroscopic measurements.
* To evaluate the safety of spectroscopic measurement of cervical tissue.

DETAILED DESCRIPTION:
If you agree to take part in this study, spectroscopic measurements on your cervix will be made for research purposes, prior to your routine colposcopy examination.

MEASUREMENT PROCEDURE:

The doctor will first place a vaginal speculum and then perform the LightTouch Ã'Â® procedure (that looks at tissue from the cervix using light). The doctor will use a fresh single use contact tube (a tube attached to the LightTouch device that helps hold it in place) and apply it gently to your cervix. This will transmit light much like a flashlight. The light will either reflect or bounce immediately off your cervix or it will enter the skin for less than a second, and then return back to the LightTouch device. Each reading will take about 5-7 minutes, and up to two readings may be taken. You may also be asked to repeat the experimental test the same day, for example 2 to 3 hours after the first test, as part of another experimental procedure to study whether the device gives the same result twice in a row on the same woman (a repeatability study). If you agree to a second (LightTouch) procedure you will again have placement of the contact tube applied gently to your cervix and another test will be taken. This could take another 5 to 7 minutes of your time.

Whether you agree to do one of the experimental tests or both of the tests, following the LightTouch experimental procedure(s), you will have a Pap smear of the endocervix (the doctor will use a small plastic brush remove cells from the endocervix canal). We will also test for human papilloma virus (HPV). HPV is a virus that is sexually transmitted is associated with abnormal Pap smears. The doctor will use two separate vials for these tests, one to take your Pap smear and the other to take more cells for an HPV test. Once the doctor takes your Pap smear and HPV test. The doctor will do the colposcopy exam using a colposcope to look at the cervix more closely to check for abnormal areas. The doctor will also apply acetic acid and Lugols if required. The doctor may also perform biopsy (remove one or more tissue samples you're your cervix) for later examination by a pathologist. If considered necessary, an ECC (Endocervical Curettage scraping of cells from the inside of the endocervix) will be performed if an abnormal area is seen.

A video image (camera) will be used to capture locations of abnormal areas and compare with the readings from the spectroscopic image. Your overall study participation time will be approximately 30 minutes. If you are asked to participate in second test and agree, it will take place directly after the first test. The spectroscopy portion in which measurements are taken takes 5 to 7 minutes to complete. If you have the second study procedure this will take an additional 15-30 minutes making your overall participation time up to 60 minutes (one hour). You may be asked to re-test one time during the same visit if the information collected is bad because of movement or if the device did not work.

The results of the LightTouch test will be compared with the results of your colposcopy and biopsy. The results of the LightTouch test test will not be used to plan your treatment. If your biopsy results show any abnormal changes, your doctor will discuss treatment options with you.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 or above
* Able to read or understand and give informed consent
* Scheduled for colposcopy
* Pap test within 120 days
* Willing to undergo a Pap test and HPV test on day of study

Exclusion Criteria:

* Pregnancy
* Menstruating on the day of colposcopy and CNDS test
* Radiation therapy to her genitourinary system within 1 year
* Prior hysterectomy
* Congenital anatomical cervical variant (e.g., double cervix)
* Friable cervix at the time of the study (i.e., a cervix that bleeds easily upon minimal contact or trauma)
* Post-coital or other significant bleeding at the time of the exam
* Excessive cervical mucous or discharge that cannot be removed and is significant enough, in the opinion of the investigator, to interfere with a Pap test or colposcopy, resulting from inflammatory, bacterial or other sources
* History of any photosensitizing disease or other disease affected by Ultra-violet radiation, (e.g., pophyria, Lupus Erythematosus).
* Undergoing phototherapy
* Recent use of photosensitizing agents, such as fluoroquinolones or retinoids).
* Patients who are pregnant are not eligible for this study.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Double-blind, Prospective, Safety-efficacy study
Sampling Method: Probability Sample
Enrollment: 1599 (Actual)
Dates: Start 2003-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Determine the efficacy of the CNDS, within the context of current ASCCP guidelines, to more effectively triage women with ASC/LSIL results, women with positive HPV results and women being followed for previous cervical dysplasia. | December 2008

SECONDARY OUTCOMES:
A second objective is to prospectively demonstrate equivalence between two versions of the CNDS used in the pivotal trial. | Q1 2009

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Flowers, MD, Principal Investigator — Emory University/Grady Hospital System
Locations (7):
- United States (7):
  - University of Arkansas, Little Rock, Arkansas
  - Orange Coast/Saddleback, Laguna Beach, California
  - Saint Francis Hospital, Hartford, Connecticut
  - University of Miami, Miami, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - University of Texas, Dallas, Texas